CLINICAL TRIAL: NCT01179347
Title: A Randomised, Double-blind, Placebo-controlled Parallel-group Trial to Confirm the Efficacy After 12 Weeks and the Safety of Tiotropium 5 Mcg Administered Once Daily Via the Respimat® Device in Patients With Cystic Fibrosis.
Brief Title: Tiotropium Bromide in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.438; 2010-019802-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

ARMS (2):
- tiotropium (Experimental): 2 inhalations once daily delivered with Respimat® inhaler
  Interventions: Drug: tiotropium Respimat® inhaler
- placebo (Placebo Comparator): 2 inhalations once daily delivered with Respimat® inhaler
  Interventions: Drug: Placebo Respimat® inhaler

INTERVENTIONS:
Drug: tiotropium Respimat® inhaler — to evaluate safety and efficacy tiotropium delivered with Respimat® inhaler compared to placebo.
  Arms: tiotropium
Drug: Placebo Respimat® inhaler — patient to receive placebo matching active drug once daily
  Arms: placebo

SUMMARY:
To date, there have been no formal clinical studies completed using tiotropium in CF patients. While there is a large body of evidence demonstrating the efficacy and safety of tiotropium in patients with Chronic Obstructive Pulmonary Disease (COPD), relatively little is known about its efficacy and safety in patients with a diagnosis of cystic fibrosis. Therefore, Boehringer Ingelheim proposed to profile the long acting anticholinergic tiotropium and to generate adequate clinical data for use as a bronchodilator in paediatric and adult CF. The phase III trial (205.438) is a part of the approved Paediatric Investigation Plan (PIP) agreed for Spiriva® Respimat® in Cystic Fibrosis.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a documented diagnosis of Cystic Fibrosis (CF) (positive sweat chloride >=60 mEq/liter, by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations.
2. Male or female patients (children less than 12 years and adolescents >12 years).
3. Patients >=5 years of age must be able to perform acceptable spirometric maneuvers, according to the American Thoracic Society (ATS) standards.
4. Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) >25% of predicted values.
5. Pre-bronchodilator FEV1 at Visit 2 must be within 15% of FEV1 at Visit 1.
6. No evidence of respiratory tract infection and no pulmonary exacerbation requiring use of intravenous/oral/inhaled antibiotics, or oral corticosteroids within 2 weeks of screening.
7. The patient or the patient's legally acceptable representative must be able to give informed consent.
8. Patients who are on a cycling TOBI® regimen must have completed at least 2 cycles every other month TOBI® administration prior to the screening visit.
9. Patients who are on daily inhaled antibiotic use must be stabilized for at least 6 weeks prior to Visit 1 (screening).
10. Patients having previously participated in study 205.339 can also be selected.

Exclusion criteria:

1. Patients with a known hypersensitivity to study drug
2. Patients who have participated in another study with an Investigational drug within one month preceding the screening visit.
3. Patients who are currently participating in another trial. Observational studies are allowed. Permission should be obtained from sponsor of other study.
4. Patients with known relevant substance abuse, including alcohol or drug abuse.
5. Adolescent and adult female patients who are pregnant or lactating, including females who have a positive serum pregnancy test at screening.
6. Female patients of child bearing potential who are not using a medically approved form of contraception.
7. Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. Patients with diabetes may participate if their disease is under good control prior to screening.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (99):
- United States (15):
  - 205.438.01004 Boehringer Ingelheim Investigational Site, Tuscon, Arizona
  - 205.438.01011 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.438.01018 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.438.01008 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.438.01014 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.438.01021 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.438.01007 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 205.438.01006 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 205.438.01001 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 205.438.01010 Boehringer Ingelheim Investigational Site, Manchester, New Hampshire
  - 205.438.01003 Boehringer Ingelheim Investigational Site, Syracuse, New York
  - 205.438.01019 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.438.01013 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.438.01005 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.438.01012 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Australia (4):
  - 205.438.61003 Boehringer Ingelheim Investigational Site, Chermside, Queensland
  - 205.438.61004 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 205.438.61001 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 205.438.61002 Boehringer Ingelheim Investigational Site, Subiaco, Western Australia
- Austria (2):
  - 205.438.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 205.438.43002 Boehringer Ingelheim Investigational Site, Salzburg
- Belgium (4):
  - 205.438.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 205.438.32004 Boehringer Ingelheim Investigational Site, Edegem
  - 205.438.32003 Boehringer Ingelheim Investigational Site, Jette
  - 205.438.32001 Boehringer Ingelheim Investigational Site, Leuven
- Canada (6):
  - 205.438.02005 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 205.438.02007 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 205.438.02004 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 205.438.02003 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 205.438.02006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 205.438.02001 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Czechia (4):
  - 205.438.42002 Boehringer Ingelheim Investigational Site, Brno
  - 205.438.42003 Boehringer Ingelheim Investigational Site, Brno
  - 205.438.42004 Boehringer Ingelheim Investigational Site, Olomouc
  - 205.438.42001 Boehringer Ingelheim Investigational Site, Prague
- France (14):
  - 205.438.33010 Boehringer Ingelheim Investigational Site, Angers
  - 205.438.33013 Boehringer Ingelheim Investigational Site, Bron
  - 205.438.33002 Boehringer Ingelheim Investigational Site, Lille
  - 205.438.33015 Boehringer Ingelheim Investigational Site, Lisieux
  - 205.438.33003 Boehringer Ingelheim Investigational Site, Montpellier
  - 205.438.33005 Boehringer Ingelheim Investigational Site, Nantes
  - 205.438.33014 Boehringer Ingelheim Investigational Site, Nice
  - 205.438.33001 Boehringer Ingelheim Investigational Site, Paris
  - 205.438.33006 Boehringer Ingelheim Investigational Site, Paris
  - 205.438.33007 Boehringer Ingelheim Investigational Site, Paris
  - 205.438.33011 Boehringer Ingelheim Investigational Site, Rennes
  - 205.438.33008 Boehringer Ingelheim Investigational Site, Roscoff
  - 205.438.33004 Boehringer Ingelheim Investigational Site, Rouen
  - 205.438.33009 Boehringer Ingelheim Investigational Site, Vannes
- Germany (9):
  - 205.438.49001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.438.49002 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.438.49012 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.438.49011 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 205.438.49006 Boehringer Ingelheim Investigational Site, Gerlingen
  - 205.438.49007 Boehringer Ingelheim Investigational Site, Giessen
  - 205.438.49005 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.438.49003 Boehringer Ingelheim Investigational Site, München
  - 205.438.49008 Boehringer Ingelheim Investigational Site, Tübingen
- Hungary (3):
  - 205.438.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 205.438.36003 Boehringer Ingelheim Investigational Site, Mosdós
  - 205.438.36004 Boehringer Ingelheim Investigational Site, Szeged
- 205.438.35301 Boehringer Ingelheim Investigational Site, Dublin, Ireland
- Israel (4):
  - 205.438.97003 Boehringer Ingelheim Investigational Site, Haifa
  - 205.438.97001 Boehringer Ingelheim Investigational Site, Jerusalem
  - 205.438.97002 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 205.438.97004 Boehringer Ingelheim Investigational Site, Tel Litwinsky
- Italy (3):
  - 205.438.39001 Boehringer Ingelheim Investigational Site, Florence
  - 205.438.39003 Boehringer Ingelheim Investigational Site, Genova
  - 205.438.39002 Boehringer Ingelheim Investigational Site, Verona
- Poland (3):
  - 205.438.48001 Boehringer Ingelheim Investigational Site, Lodz
  - 205.438.48002 Boehringer Ingelheim Investigational Site, Rabka-Zdrój
  - 205.438.48003 Boehringer Ingelheim Investigational Site, Warsaw
- Portugal (4):
  - 205.438.35001 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.438.35002 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.438.35003 Boehringer Ingelheim Investigational Site, Porto
  - 205.438.35004 Boehringer Ingelheim Investigational Site, Porto
- Russia (5):
  - 205.438.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 205.438.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 205.438.07003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.438.07004 Boehringer Ingelheim Investigational Site, Voronezh
  - 205.438.07002 Boehringer Ingelheim Investigational Site, Yaroslavl
- Slovakia (3):
  - 205.438.42102 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 205.438.42101 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.438.42103 Boehringer Ingelheim Investigational Site, Košice
- 205.438.27001 Boehringer Ingelheim Investigational Site, Cape Town, South Africa
- Spain (4):
  - 205.438.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 205.438.34001 Boehringer Ingelheim Investigational Site, Madrid
  - 205.438.34002 Boehringer Ingelheim Investigational Site, Madrid
  - 205.438.34004 Boehringer Ingelheim Investigational Site, Valencia
- Switzerland (4):
  - 205.438.41003 Boehringer Ingelheim Investigational Site, Basel
  - 205.438.41004 Boehringer Ingelheim Investigational Site, Bern
  - 205.438.41001 Boehringer Ingelheim Investigational Site, Zurich
  - 205.438.41002 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (6):
  - 205.438.44009 Boehringer Ingelheim Investigational Site, Brighton
  - 205.438.44007 Boehringer Ingelheim Investigational Site, Cambridge
  - 205.438.44004 Boehringer Ingelheim Investigational Site, Leeds
  - 205.438.44005 Boehringer Ingelheim Investigational Site, Nottingham
  - 205.438.44002 Boehringer Ingelheim Investigational Site, Plymouth
  - 205.438.44003 Boehringer Ingelheim Investigational Site, Sheffield

REFERENCES:
- [Derived] Ratjen F, Koker P, Geller DE, Langellier-Cocteaux B, Le Maulf F, Kattenbeck S, Moroni-Zentgraf P, Elborn JS; Tiotropium Cystic Fibrosis Study Group. Tiotropium Respimat in cystic fibrosis: Phase 3 and Pooled phase 2/3 randomized trials. J Cyst Fibros. 2015 Sep;14(5):608-14. doi: 10.1016/j.jcf.2015.03.004. Epub 2015 Mar 26. PMID 25819269
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/205/205.438_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First part: double-blind, duration was 12 weeks, 464 patients were randomised to either Tio R5 or placebo in a 2:1 ratio, but 1 randomised patient was not treated. Second part: open-label, all patients received the active treatment for a minimum of 12 weeks to enlarge the safety database.
Groups:
- Placebo: Matching Placebo once daily (qd) delivered by the Respimat inhaler as add-on therapy to usual care in patients with cystic fibrosis.
- Tio R5 qd: Tiotropium 5 mcg qd delivered by the Respimat inhaler as add-on therapy to usual care in patients with cystic fibrosis.
Period: Double-blind Period (12 Weeks)
Arm/Group | Placebo | Tio R5 qd
Started | 155 (Entered and treated in double-blind period.) | 308 (Entered and treated in double-blind period.)
Completed | 147 (Completed double-blind period.) | 294 (Completed double-blind period.)
Not Completed | 8 | 14
Not completed — Adverse Event | 2 | 6
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 2 | 4
Period: Open-label Period (12 Weeks)
Arm/Group | Placebo | Tio R5 qd
Started | 147 (Treated in open-label period.) | 294 (Treated in open-label period.)
Completed | 132 (Completed open-label period.) | 278 (Completed open-label period.)
Not Completed | 15 | 16
Not completed — Adverse Event | 5 | 9
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tio R5 qd | Total
Number analyzed (Participants) | 155 | 308 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.6 (13.6) | 19.3 (12.0) | 19.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 139 | 204
  Male | 90 | 169 | 259

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve 0-4 Hours (AUC0-4h) Response
Description: Mixed Model Repeated Measurement (MMRM) results. Response was defined as change from baseline in percent of predicted at the end of 12-week double-blind treatment period and is therefore expressed in percent of predicted. Means are adjusted for treatment, visit, treatment-by-visit interaction, age group (<= 11, >=12), baseline and baseline-by-visit interaction. FEV1 AUC0-4h was normalised for time and was calculated using the trapezoidal rule divided by the observation time (4 h).
Time Frame: 30 minutes (min) before first dosing of study drug (defined as baseline), at 1 hour (h), 2 h , 3 h, and 4 h post dosing at day 1 and at 30 min before dosing, at 1 hour, 2 h , 3 h, and 4 h post dosing after 12 weeks.
Population: Full Analysis Set (FAS) with imputation reduced to patients with observed wash-out compliance. The FAS was defined as all patients in the treated set who had at least 1 baseline pulmonary function test (PFT) measurement and at least 1 post-baseline on-treatment PFT measurement. No patients <5 years of age were included in the FAS.
Measure: Mean (Standard Error); unit: Percent of predicted
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 146 | 292
Percent of predicted | 0.87 (0.80) | 2.51 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Hierarchical testing procedure was applied for both co-primary endpoints to maintain the overall alpha level. If and only if statistical superiority of the Tio R5 qd compared to Placebo in FEV1 AUC0-4h was demonstrated at the 1 sided alpha level of 0.025, confirmatory comparison in the second co-primary endpoint, at the same alpha level of 0.025 could be done; Test type: Superiority or Other; p = 0.092, Mixed Models Analysis — Two-sided p-value; Restricted maximum likelihood (REML)-based MMRM. Adjusted for treatment, visit, treatment-by-visit, age group, baseline and baseline-by-visit; Mean Difference (Final Values) = 1.64, 95% CI [-0.27 to 3.55], Standard Error of Mean 0.97 — Tio R5 qd minus Placebo

2. Primary Outcome: Trough FEV1 Response
Description: MMRM results. Response was defined as change from baseline in percent of predicted at the end of 12-week double-blind treatment period and is therefore expressed in percent of predicted. Trough FEV1 was defined as the pre-dose FEV1 measured just prior to the administration of randomised treatment. Means are adjusted for treatment, visit, treatment-by-visit interaction, age group (<= 11, >=12), baseline and baseline-by-visit interaction.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of predicted
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 144 | 287
Percent of predicted | 0.72 (0.80) | 2.12 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Hierarchical testing for co-primary endpoints, confirmatory only if previous hypotheses had been successful,; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis — Two-sided p-value; REML-based MMRM. Adjusted for treatment, visit, treatment-by-visit, age group, baseline and baseline-by-visit; Mean Difference (Final Values) = 1.40, 95% CI [-0.50 to 3.30], Standard Error of Mean 0.97 — Tio R5 qd minus Placebo

3. Secondary Outcome: Forced Vital Capacity (FVC) Area Under the Curve 0-4 Hours (AUC0-4h) Response
Description: MMRM results. Response was defined as change from baseline in percent of predicted at the end of 12-week double-blind treatment period and is therefore expressed in percent of predicted. Means are adjusted for treatment, visit, treatment-by-visit interaction, age group (<= 11, >=12), baseline and baseline-by-visit interaction. FVC AUC0-4h was normalised for time and was calculated using the trapezoidal rule divided by the observation time (4 h).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of predicted
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 137 | 282
Percent of predicted | 0.17 (0.75) | 1.27 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis — Two-sided p-value; REML-based MMRM. Adjusted for treatment, visit, treatment-by-visit, age group, baseline and baseline-by-visit; Mean Difference (Final Values) = 1.09, 95% CI [-0.68 to 2.86], Standard Error of Mean 0.90 — Tio R5 qd minus Placebo

4. Secondary Outcome: Trough FVC Response
Description: MMRM results. Response was defined as change from baseline in percent of predicted at the end of 12-week double-blind treatment period and is therefore expressed in percent of predicted. Trough FCV was defined as the pre-dose FVC measured just prior to the administration of randomised treatment. Means are adjusted for treatment, visit, treatment-by-visit interaction, age group (<= 11, >=12), baseline and baseline-by-visit interaction.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of predicted
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 135 | 277
Percent of predicted | 0.30 (0.77) | 1.51 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis — Two-sided p-value; REML-based MMRM. Adjusted for treatment, visit, treatment-by-visit, age group, baseline and baseline-by-visit; Mean Difference (Final Values) = 1.20, 95% CI [-0.62 to 3.02], Standard Error of Mean 0.93 — Tio R5 qd minus Placebo

5. Secondary Outcome: Pre-bronchodilator Forced Expiratory Flow Between 25 Percent and 75 Percent of the FVC (FEF25-75) Response
Description: MMRM results. Response was defined as change from baseline in percent of predicted at the end of 12-week double-blind treatment period and is therefore expressed in percent of predicted. FEF25-75 is also known as maximum mid-expiratory flow and was measured before bronchodilator (salbutamol) use. Means are adjusted for treatment, visit, treatment-by-visit interaction, age group (<= 11, >=12), baseline and baseline-by-visit interaction.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of predicted
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 135 | 277
Percent of predicted | 2.15 (1.48) | 3.02 (1.05)
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.62, Mixed Models Analysis — Two-sided p-value; REML-based MMRM. Adjusted for treatment, visit, treatment-by-visit, age group, baseline and baseline-by-visit; Mean Difference (Final Values) = 0.86, 95% CI [-2.59 to 4.32], Standard Error of Mean 1.76 — Tio R5 qd minus Placebo

6. Secondary Outcome: Percentage of Participants With at Least 1 Pulmonary Exacerbation During Double-blind Treatment
Description: Selected questions from the Respiratory and Systemic Symptoms Questionnaire (RSSQ), the investigator assessment of physical findings and pulmonary function, and the use of intravenous antibiotics as a concomitant therapy were used to determine if a cystic fibrosis-related pulmonary exacerbation had occurred.
Time Frame: 12 weeks
Population: FAS reduced to patients having RSSQ information on day 29, 57 or 85.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 102 | 214
Percentage of Participants | 7.8 | 8.9
Statistical Analysis 1: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.84, Regression, Logistic — Two-sided p-value; Adjusted for treatment, age group, baseline weight and baseline FEV1 percent predicted; Odds Ratio (OR) = 1.092, 95% CI [0.453 to 2.633] — Tio R5 qd versus Placebo

7. Secondary Outcome: Change From Baseline in Revised Cystic Fibrosis Questionnaire (CFQ-R) Score
Description: Different format of CFQ-R are used depending of the patients' age. Adolescent and adult format of CFQ-R is used for patients of 14 years and older, for younger children a parent version and a children format is used. In case parent and children questionnaires were filled out, the children questionnaire is taken into account. Scores were calculated for each domain of the CFQ-R which are presented separately. A score of 100 corresponds to the highest quality of life possible, whereas a score of 0 corresponds to the lowest quality of life possible. Increasing score indicates better health.
Time Frame: Baseline and 12 weeks
Population: FAS reduced to patients having CFQ-R information at baseline and at week 12.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tio R5 qd
Number analyzed (Participants) | 130 | 255
Units on a scale
  Adolescents: Physical (N=83, N=162) | -0.85 (14.40) | -0.15 (12.95)
  Adolescents: Role (N=78, N=157) | 0.85 (12.99) | -0.42 (13.30)
  Adolescents: Vitality (N=82, N=161) | -1.22 (18.06) | 0.05 (14.08)
  Adolescents: Emotion (N=82, N=161) | -1.54 (12.05) | -0.99 (12.96)
  Adolescents: Social (N=82, N=159) | -1.69 (10.09) | 0.70 (10.19)
  Adolescents: Body Image (N=82, N=159) | 0.14 (16.14) | 3.14 (15.11)
  Adolescents: Eating (N=82, N=161) | -1.49 (14.89) | 1.38 (10.74)
  Adolescents: Treatment burden (N=82, N=160) | 0.95 (14.73) | 0.56 (14.84)
  Adolescents: Health perseptions (N=82, N=159) | -0.81 (13.83) | 0.77 (16.68)
  Adolescents: Weight (N=80, N=160) | -2.08 (29.22) | 3.75 (26.96)
  Adolescents: Respiratory (N=80, N=159) | 0.97 (13.83) | -0.77 (15.19)
  Adolescents: Digestion (N=80, N=159) | -0.83 (17.03) | 0.49 (12.40)
  Children: Physical (N=47, N=93) | -2.84 (15.67) | 1.43 (15.19)
  Children: Social (N=46, N=93) | 2.80 (15.73) | 1.59 (15.70)
  Children: Body Image (N=46, N=93) | -1.21 (18.48) | 4.66 (25.71)
  Children: Emotion (N=47, N=93) | -1.24 (12.83) | 1.12 (12.18)
  Children: Eating (N=47, N=93) | 2.84 (19.03) | 0.72 (20.18)
  Children: Treatment burden (N=46, N=93) | 0.72 (15.43) | -0.48 (19.10)
  Children: Respiratory (N=46, N=93) | -0.91 (15.34) | -1.61 (16.81)
  Children: Digestion (N=46, N=92) | 2.17 (22.66) | -1.09 (29.84)

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 30 days after last administration of trial drug, for AE analyses over open-label period and over the study. Over the double-blind period, 30 days of wash-out is only used for premature discontinued patients.
Arm/Group | Placebo Randomized Group Over the Double-Blind Period | Tio 5mcg Randomized Group Over the Double-Blind Period | Placebo Randomized Group Over the Open-Label Period | Tio 5mcg Randomized Group Over the Study
Serious Adverse Events (participants affected / at risk) | 13/155 | 36/308 | 24/147 | 62/308
Other Adverse Events (participants affected / at risk) | 27/155 | 63/308 | 56/147 | 186/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Randomized Group Over the Double-Blind Period (N=155) | Tio 5mcg Randomized Group Over the Double-Blind Period (N=308) | Placebo Randomized Group Over the Open-Label Period (N=147) | Tio 5mcg Randomized Group Over the Study (N=308)
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Cystic fibrosis (Congenital, familial and genetic disorders) | 2 | 6 | 7 | 11
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 | 2 | 3 | 2
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 2
Device occlusion (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 3 | 6
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 2
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 4 | 3 | 10
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 5 | 1 | 6
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Bacterial test positive (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Forced expiratory volume decreased (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 9
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Antibiotic prophylaxis (Surgical and medical procedures) | 1 | 0 | 0 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 0 | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Randomized Group Over the Double-Blind Period (N=155) | Tio 5mcg Randomized Group Over the Double-Blind Period (N=308) | Placebo Randomized Group Over the Open-Label Period (N=147) | Tio 5mcg Randomized Group Over the Study (N=308)
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 19
Nausea (Gastrointestinal disorders) | 0 | 0 | 8 | 0
Pyrexia (General disorders) | 10 | 15 | 13 | 28
Bronchitis (Infections and infestations) | 0 | 0 | 10 | 22
Nasopharyngitis (Infections and infestations) | 0 | 0 | 11 | 25
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 18
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 24
Headache (Nervous system disorders) | 0 | 0 | 8 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 55 | 30 | 80
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 16
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.